CLINICAL TRIAL: NCT02644603
Title: Safety and Efficacy of the Enhanced Recovery After Surgery(ERAS) After Liver Resection for Primary Liver Cancer: a Multicenter, Randomized, Controlled Clinical Study
Brief Title: Effect of Enhanced Recovery After Surgery(ERAS) After Liver Resection for Primary Liver Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other); RenJi Hospital (Other); Anhui Provincial Hospital (Other Government); Subei People's Hospital of Jiangsu Province (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-ERAS-MRCT-1511
Record Dates: First submitted 2015-12-15; First posted 2016-01-01 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Enhanced Recovery After Surgery; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Recovery After Surgery (Experimental): Patients underwent ERAS protocol
  Interventions: Procedure: Enhanced Recovery After Surgery
- Conventional Treatment (No Intervention): Patients underwent conventional treatment

INTERVENTIONS:
Procedure: Enhanced Recovery After Surgery — Before operation:
  Preoperative optimization of organ function, No preoperative bowel preparation, Prohibit eating 6h, drinking water 2h before operation, Oral rehydration before operation.
  In operation:
  Optimized combined anesthesia, Minimal invasive operations, Normothermia, Minimal use of tubes and drains.
  After operation:
  Postoperative analgesia and antiemetic, Early mobilization, Oral nutrition, Early and scheduled mobilization.
  Other Names: Fast Track Surgery
  Arms: Enhanced Recovery After Surgery

SUMMARY:
The purpose of this study is to evaluate Enhanced Recovery After Surgery(ERAS) protocol versus conventional treatment on patients who underwent liver resection for hepatocellular carcinoma(HCC).

DETAILED DESCRIPTION:
212 patients are randomly recruited from inpatients of Shanghai Zhongshan Hospital, Eastern Hepatobiliary Surgery Hospital, RenJi Hospital, Anhui Provincial Hospital, Subei People's Hospital of Jiangsu Province and Affiliated Tumor Hospital of Nantong University from February 2016 to July 2016. Randomly assigned about half of the patients to receive Enhanced Recovery After Surgery(ERAS) protocol and the other half to receive conventional treatment. Evaluate the safety and efficacy of the ERAS protocol.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HCC with indications for surgery
* Without any surgical contraindications
* Under went open liver resection
* Operation ranges less than 4 hepatic segments
* Informed consent

Exclusion Criteria:

* Not suitable for surgery
* Benign lesions or other lesions proved by pathology
* Surgical procedure changed during operation or combined evisceration
* Refused to participate or drop out

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Treatment related complications | Up to 1 month since operation
  Number of adverse events that are related to treatment of each patients, and hospital readmission

SECONDARY OUTCOMES:
Length of stay in hospital | From the day a patient be hospitalized to the day discharged, up to 1 month.
  Length of stay in hospital (days)
Total hospitalization costs | From the day a patient be hospitalized to the day discharged, up to 1 month.
  Total hospitalization costs (RMB yuan).
Preoperative and postoperative body weight | One day before operation, and the day patient discharged, up to 1 month.
  Patient's body weight in kg.
Hemoglobin (Hb) test Hb/ALB/PRE-A(g/L), | Day before operation and day 1/3/5 after operation.
  Hb in g/L.
Albumin (ALB) | Day before operation and day 1/3/5 after operation.
  ALB in g/L.
PRE-Albumin (PRE-A) | Day before operation and day 1/3/5 after operation.
  PRE-A in g/L
International Normalized Ratio (INR) | Day before operation and day 1/3/5 after operation.
  INR in seconds.
Platelet (PLT) | Day before operation and day 1/3/5 after operation.
  PLT in 10^9/L
Blood Urea Nitrogen (BUN) | Day before operation and day 1/3/5 after operation.
  BUN in mmol/L
Blood Creatinine (sCr) | Day before operation and day 1/3/5 after operation.
  sCr in umol/L
Alanine Transferase (ALT) | Day before operation and day 1/3/5 after operation.
  ALT in U/L
Aspartate Transaminase (AST) | Day before operation and day 1/3/5 after operation.
  AST in U/L
Interleukin-6 (IL-6) | Day before operation and day 1/3/5 after operation.
  IL-6 in (pg/ml)
Interferon (IFN-γ) | Day before operation and day 1/3/5 after operation.
  IFN-γin pg/ml.
Tumor necrosis factor-α (TNF-α) | Day before operation and day 1/3/5 after operation.
  TNF-αin pg/ml
Serum complement | Day before operation and day 1/3/5 after operation.
  C3 and C4 in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, MD, PhD, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sun HC, Qin LX, Lu L, Wang L, Ye QH, Ren N, Fan J, Tang ZY. Randomized clinical trial of the effects of abdominal drainage after elective hepatectomy using the crushing clamp method. Br J Surg. 2006 Apr;93(4):422-6. doi: 10.1002/bjs.5260. PMID 16491462
- [Background] Wilmore DW, Kehlet H. Management of patients in fast track surgery. BMJ. 2001 Feb 24;322(7284):473-6. doi: 10.1136/bmj.322.7284.473. No abstract available. PMID 11222424
- [Background] Ni CY, Yang Y, Chang YQ, Cai H, Xu B, Yang F, Lau WY, Wang ZH, Zhou WP. Fast-track surgery improves postoperative recovery in patients undergoing partial hepatectomy for primary liver cancer: A prospective randomized controlled trial. Eur J Surg Oncol. 2013 Jun;39(6):542-7. doi: 10.1016/j.ejso.2013.03.013. Epub 2013 Apr 4. PMID 23562361